CLINICAL TRIAL: NCT00969462
Title: Association Between Response to Aggressive Chemotherapy and Doxorubicin Pharmacokinetics in Non Hodgkin's Lymphoma Patients
Brief Title: Doxorubicin Pharmacokinetics and Response in Non Hodgkin's Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1. NHL; non
Record Dates: First submitted 2009-08-17; First posted 2009-09-01 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2012-03

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Doxorubicin; pharmacokinetics; non-Hodgkin's lymphoma; response; association between response to chemotherapy; myelosuppression degree; doxorubicin pharmacokinetics
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxorubicin (No Intervention): Single arm
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin — measurements of serum Doxorubicin levels

SUMMARY:
In previous studies, the investigators found that in patients with Hodgkin's lymphoma (HL) treated with ABVD (adriamycin, bleomycin, vinblastine and decarbazine) the absence of alopecia may predict for a poor response to treatment [complete remission (CR) rate 79% versus 31%, P < 0.0005, respectively]. Also, patients without alopecia had fewer episodes of either leucopenia, neutropenia, deferral of treatment courses or number of courses with dose reduction [88% vs. 62.5%, P=0.05, for the presence of at least one of them].

One of the explanations for this phenomenon is related to a lower systemic exposure of chemotherapeutic drugs in patients who retain their hair. There is a wide interpatient variability in the pharmacokinetic and pharmacodynamic parameters of doxorubicin systemic exposure and the degree of myelosuppression.

In a pilot study on 18 patients the investigators could not find the previous association between alopecia, response to chemotherapy and bone marrow depression. However, when analyzing doxorubicin pharmacokinetics, patients who had no remission had 2 fold lower AUC (area under the curve) and 3 fold lower peaks (p=0.06). The investigators' lack to approve the previous findings might be explained by the small study group.

DETAILED DESCRIPTION:
Aim of the study:

To evaluate the association between response to chemotherapy, the degree of myelosuppression and the pharmacokinetics of doxorubicin in non-Hodgkin's lymphoma (NHL) patients.

Methods:

Study protocol:

1. At diagnosis

   Demographic and clinical parameters be collected (Appendix 1)
2. At course 2:

1. Doxorubicin will be given by 5-7 minutes infusion before the other medications (Doxorubicin doses will be collected (Appendix 1))

2. Blood will be sampled in course 2, at:

0 minutes 30 minutes 120 minutes 24 hours

Two 2ml EDT tubes will be drawn at each time The tubes will be centrifuged at 3000 RPM for 15 min. Plasma samples will be stored in - 700C

3. At the end of chemotherapy courses the following data will be collected (Appendix 2):

1. Episodes of bone marrow depression (leucopenia, neutropenia) Treatment delays Dose reductions Neutropenic fever
2. Remission status

[Complete remission (CR) - disappearance of clinical signs and symptoms of NHL along with normal laboratory and radiological findings].

4. At the end of one year of CR

Remission status

Number of patients: 30

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Biopsy proven intermediate grade NHL
* No previous chemotherapy
* At least 4 courses of R-CHOP at maximal doses are planned
* An informed consent

Exclusion Criteria:

* Do not meet all inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Doxorubicin, pharmacokinetics at first chemotherapy course | 1 year

SECONDARY OUTCOMES:
Association between doxorubicin pharmacokinetics and response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Avishay Elis, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Departmetn of Medicine. Meir Medical Center, Kfar Saba, Israel